CLINICAL TRIAL: NCT05520125
Title: Treatment of Patients With Segmental Bone Tissue Defects Using Mesenchymal Stem Cells Enriched by Extracellular Vesicles
Brief Title: Treatment of Patients With Bone Tissue Defects Using Mesenchymal Stem Cells Enriched by Extracellular Vesicles
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus (Other Government)
Collaborators: Belarusian Medical Academy of Post-Graduate Education (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBCE_MSCVesicles
Record Dates: First submitted 2022-08-26; First posted 2022-08-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Segmental Fracture - Bone Loss
Keywords: bone defects, mesenchymal stem cells, extracellular vesicles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with bone defects receiving standard treatment and MSC enriched with extracellular vesicles (Experimental): Patients with bone defects receiving standard treatment and MSC enriched with extracellular vesicles
  Interventions: Biological: Mesenchymal stem cells enriched by extracellular vesicles; Other: Standard treatment of bone defects
- Patients with bone defects receiving standard treatment (Active Comparator): Patients with bone defects receiving standard surgical treatment
  Interventions: Other: Standard treatment of bone defects

INTERVENTIONS:
Biological: Mesenchymal stem cells enriched by extracellular vesicles — Mesenchymal stem cells enriched by extracellular vesicles
  Arms: Patients with bone defects receiving standard treatment and MSC enriched with extracellular vesicles
Other: Standard treatment of bone defects — Standard surgical treatment of bone defects

SUMMARY:
Treatment of patients with segmental bone tissue defects using mesenchymal stem cells enriched by extracellular vesicles

DETAILED DESCRIPTION:
The aims of the project are to develop a technology for obtaining mesenchymal stem cells extracellular vesicles; to develop biomedical cell product based on mesenchymal stem cells enriched with own extracellular vesicles; to conduct the clinical trials of the biomedical cell product in the treatment of patients with segmental bone tissue defects

ELIGIBILITY:
Inclusion Criteria:

* age 18-50 years;
* non-union fractures of the tubular bones of the upper limb;
* segmental defects of the bone tissue of the tubular bones of the upper limbs;
* absence of severe comorbidity worsening the patient's prognosis.

Exclusion Criteria:

* pregnancy;
* acute inflammatory processes;
* viral hepatitis B and C, HIV infection, syphilis and other viral and bacterial infections;
* autoimmune diseases;
* allergic reactions in the acute stage, established hypersensitivity to any component of the biomedical cell product;
* mental and behavioral disorders that make it impossible for patients to participate in the study, drug and/or alcohol addiction;
* patients with malignant tumors including a history.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse effects associated with the therapy | 1 year
  Determination of adverse effects associated with the therapy
Adverse effects associated with the therapy | 1 month
  Determination of adverse effects associated with the therapy
Percent of completely recovered patients with segmental bone tissue defects | 1 year
  Percent of completely recovered patients with segmental bone tissue defects

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Hancharou, Dr, Study Chair — Institute for biophysics and cellular engineering NAS of Belarus
Locations (1):
- Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: No